CLINICAL TRIAL: NCT05334277
Title: FurmOnertinib Mesylate With or Without Chemotherapy +/- bevacizUmab as firSt Line Treatment in Advanced Non-small Cell Lung Cancer Patients With Uncleared Epidermal Growth Factor Receptor (EGFR) Mutation Positive Circulating Tumor Cell DNA
Brief Title: Furmonertinib Monotherapy and Combination Therapy in Advanced EGFR Mutant NSCLC With Uncleared ctDNA
Acronym: FOCUS-C
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Allist Pharmaceuticals, Inc. (Industry); GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-296-01
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Furmonertinib 80mg QD (Experimental): Furmonertinib (AST2818) 80mg QD. All patients enrolled into this group will receive furmonertinib 80mg daily.
  Interventions: Drug: Furmonertinib
- Group B1: Furmonertinib 80mg QD (Experimental): Furmonertinib (AST2818) 80mg QD. All patients enrolled into this group will receive furmonertinib 80mg daily.
  Interventions: Drug: Furmonertinib
- Group B2: Furmonertinib plus chemotherapy (Experimental): Furmonertinib 80 mg QD and platinum-based chemotherapy All patients enrolled into this group will receive furmonertinib 80 mg daily, in combination with Pemetrexed (500 mg/m2) plus carboplatin (AUC 5) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Interventions: Drug: Furmonertinib/Pemetrexed/Carboplatin
- Group B3: Furmonertinib plus chemotherapy and bevacizumab (Experimental): Furmonertinib 80 mg QD plus platinum-based chemotherapy and bevacizumab All patients enrolled into this group will receive furmonertinib 80 mg daily, in combination with Pemetrexed (500 mg/m2) plus carboplatin (AUC 5) plus bevacizumab (7.5mg/kg) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by pemetrexed (500 mg/m2) with bevacizumab (7.5mg/kg) maintenance every 3 weeks.
  Interventions: Drug: Furmonertinib/Pemetrexed/Carboplatin/Bevacizumab

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80mg QD
  Other Names: AST2818
  Arms: Group A: Furmonertinib 80mg QD
Drug: Furmonertinib — Furmonertinib 80mg QD
  Other Names: AST2818
  Arms: Group B1: Furmonertinib 80mg QD
Drug: Furmonertinib/Pemetrexed/Carboplatin — Furmonertinib 80mg daily + Pemetrexed (500 mg/m2) plus carboplatin (AUC 5) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Arms: Group B2: Furmonertinib plus chemotherapy
Drug: Furmonertinib/Pemetrexed/Carboplatin/Bevacizumab — Furmonertinib 80mg daily + Pemetrexed (500 mg/m2) plus carboplatin (AUC 5) plus bevacizumab (7.5mg/kg) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by pemetrexed (500 mg/m2) with bevacizumab (7.5mg/kg) maintenance every 3 weeks.
  Arms: Group B3: Furmonertinib plus chemotherapy and bevacizumab

SUMMARY:
EGFR mutation positive advanced NSCLC patients with uncleared ctDNA have poor prognosis, whether they can benefit from combination therapy has not been reported. This study aims to investigate the efficacy and safety of combination therapy compared with furmonertinib monotherapy in advanced EGFR mutant NSCLC with uncleared circulating tumor cell DNA.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open label, clinical study in China.

In total the study aims to screen 720 patients and enroll approximately 280 advanced NSCLC patients with EGFR mutation positive circulating tumor cell DNA, consisting of 47 patients whose ctDNA is cleared after 3 weeks furmonertinib will receive furmonertinib monotherapy, and approximately 233 patients with uncleared ctDNA after 3weeks furmonertinib monotherapy will receive furmonertinib alone or furmonertinib in combination with chemotherapy or furmonertinib in combination with chemotherapy and bevacizumab in the main trial. In the main part of the trial, for the approximately 233 patients with uncleared ctDNA, there are 2 / 2 / 1 in 5 chances of receiving furmonertinib alone, furmonertinib plus chemotherapy, or furmonertinib plus chemotherapy and bevacizumab. The treatment is decided at random by a computer.

The study involves a Screening Period, Induction treatment period, Treatment Period, and Follow up Period. Whilst receiving study medication, it is expected patients will attend, on average, approximately 9 visits. Each visit will last about 2 to 6 hours depending on the arrangement of medical assessments by the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to any study specific procedures;
2. at least 18 years of age;
3. ECOG PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks, life expectancy ≥12 weeks;
4. Pathologically confirmed non-squamous Non-Small Cell Lung Cancer (NSCLC);
5. Locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy;
6. Patient with EGFR 19Del or L858R mutation diagnosed histologically or cytologically and confirmed by ctDNA, the reports must be issued or recognized by Tier 3A hospitals. The mutations above may exist alone or together;
7. Patients must have untreated advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy;
8. According to RECIST 1.1, patients have at least one tumor lesion at baseline that meets the following requirements: accurately and repeatably measurable at baseline;
9. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the first dose, and the pregnancy test (blood or urine test) must be negative; female subjects must not be lactating;
10. Willing to use contraception as appropriate during the study and for a period after discontinuing study treatment;
11. Voluntary and agree to follow the study treatment protocol as well as follow-up plan, and can accept the oral medicine treatment;
12. Voluntary and agree to sign the informed consent for genetic research, and provide enough fresh blood samples for central NGS testing.

Exclusion Criteria:

1. squamous cell lung carcinoma;
2. History of hypersensitivity to active or inactive excipients of investigational product (IP) or drugs with a similar chemical structure or class to investigational product (IP);
3. Confirmed EGFR 20 exon insertion mutations at any time after the initial diagnosis;
4. Patient who receive prior treatment including any of the following:

   * Any Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI);
   * The patients who have received intrapleural perfusion therapy can only be enrolled 28 days or more after the pleural effusion is stable;
   * Major surgery within 4 weeks of the first dose of investigational product (IP);
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP;
   * CYP3A4 strong inhibitor or strong inducer is used within 7 days prior to the first dose, or need to receive these drugs during the study period;
   * Traditional Chinese medicine and traditional Chinese medicine preparations with anti-tumor as indications and with adjuvant treatment of tumor is used within 7 days prior to the first dose, or need to receive these drugs during the study period;
   * Patients who are receiving drugs known to prolong QTc interval or may cause torsade de pointe and need to continue to receive these drugs during the study period;
   * The time from the treatment with any other investigational product or its analogue to the first dose does not exceed 5 half-lives of the drug or 14 days, whichever is longer;
5. Prior treatment with any systemic anti-cancer therapy for advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiation including chemotherapy, biologic therapy, target therapy, immunotherapy, or any investigational drug, except neoadjuvant or adjuvant therapy before 6 months prior to the first dose;
6. At the beginning of study treatment, any unresolved toxic reaction to prior treatment is present, which exceeds Grade 1 in accordance with Common Terminology Criteria for Adverse Events (CTCAE) (except for alopecia), and exceeds Grade 2 for prior platinum treatment-related neuropathy.
7. Spinal cord compression; symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids.
8. Diagnosed other malignant tumors or had a history of other malignant tumors in last 5 years, except for skin basal cell carcinoma, cervical carcinoma in situ and breast ductal carcinoma in situ which have been effectively controlled;
9. Recent active digestive diseases such as duodenal ulcer, ulcerative colitis, ileitis, intestinal perforation, intestinal fistula, or other conditions that may cause gastrointestinal bleeding or perforation as the researchers may prescribe. Or refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of IP;
10. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, and active infection, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial;
11. Past medical history of Interstitial Lung Disease (ILD), drug-induced Interstitial Lung Disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active Interstitial Lung Disease;
12. Any evidence of known corneal injury;
13. Inadequate bone marrow reserve or organ function;
14. QT prolongation or any clinically important abnormalities in rhythm or heart function;
15. Patients who may have poor compliance with the research procedures and requirements, etc., as judged by investigators;
16. Pregnancy or lactation;
17. Patients who have had allogeneic bone marrow transplantation or received blood transfusion within 120 days prior to genetic sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The primary analysis of Progression-free survival (PFS) based on investigator assessment will occur when PFS maturity is observed at approximately 34 months after the first patient begin study treatment
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable Response Evaluation Criteria in Solid Tumors (RECIST) assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Analysis will occur when PFS maturity is observed at approximately 34 months from the first patient begin study treatment
  Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments) is defined as the number (%) of patients with response
Disease Control Rate (DCR) | Analysis will occur when PFS maturity is observed at approximately 34 months from the first patient begin study treatment
  Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator.
Duration of Response (DoR) | Duration of Response analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 34 months from the first patient begin study treatment
  Duration of Response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Overall Survival (OS) | The analysis of OS will be conducted at 2 time points: when PFS maturity is observed at approximately 34 months after the first patient begin study treatment, and when OS maturity is observed at approximately 70 months after the first patient begin study
  Overall survival is defined as the time from beginning of study treatment until death due to any cause.
Landmark Overall Survival (LOS) | The analysis of Landmark Overall Survival will be conducted at 2 time points: when PFS maturity is observed at approximately 34 months after the first patient begin study treatment, and when Overall Survival maturity is observed at approximately 70 month
  Landmark Overall Survival at 1, 3 and 5 years will look at the number of patients alive at 1-, 3- and 5-year time points.
Adverse Events | From the start of study drug to 30 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0.

OTHER OUTCOMES:
Change from baseline and time to deterioration in gene mutation spectrum of ctDNA | Gene mutation spectrum changes based on ctDNA analysis will occur when PFS maturity is observed at approximately 34 months from the first patient begin study treatment
  Gene mutation spectrum of ctDNA will be detected by NGS. The development of resistance will be monitored.
Circulating tumor DNA (ctDNA) clearance rate | The data of ctDNA clearance rate will be collected at 2 time points: 3 weeks following the first dose of study drug in induction treatment, and 3 weeks after randomization
  The proportion of patients with circulating tumor DNA clearance after 3 weeks study treatment.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - The First Hospital of Jilin University, Changchun
  - Sichuan Provincial People's Hospital, Chengdu
  - Dongguan People's Hospital, Dongguan
  - Affiliated Dongyang Hospital of Wenzhou Medical University, Dongyang People's hospital, Dongyang
  - The First People's Hospital of Foshan, Foshan
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yat-sen University cancer center, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou
  - Jiangmen Central Hospital, Affiliated Jiangmen Hospital of Sun Yat-sen University, Jiangmen
  - Affiliated Jinhua Hospital, Zhejiang University School of Medicine, Jinhua
  - Mianyang Central Hospital, Mianyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital & Institute, Shenyang
  - Shijiazhuang People's hospital, Shijiazhuang
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - The Third Affiliated Hospital of Wenzhou Medical University, Rui'an People's Hospital, Wenzhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Yijishan Hospital, Wannan Medical College, Wuhu
  - Tangdu Hospital, Fourth Military Medical University, Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No